CLINICAL TRIAL: NCT04883502
Title: Study of the Role of the Induced Membrane in the Reconstruction of Bone Loss in the Limbs
Acronym: MEMBRAN
Status: Recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PPRC03; 2021-A00561-40 (Other: IDRCB)
Record Dates: First submitted 2021-04-28; First posted 2021-05-12 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Bone Loss
Keywords: Masquelet technique; Induced membrane technique
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 1 blood sample
  * 3 fragments of induced membrane
  * 1 fragment of periosteum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood sample collection — A blood sample will be collected at enrollment.
Biological: Other biological sample collection — The following biological samples will be collected during the first surgery:
  * 1 blood sample
  * 3 fragments of induced membrane
  * 1 fragment of periosteum
Diagnostic Test: Surgical waste collection — The pieces of polymethylmethacrylate surgical cement will be collected during the second surgery.
Diagnostic Test: Radiological examination and functional exploration — A radiological examination and a functional exploration will be performed 6 weeks, 3 months and 6 months after the first surgery

SUMMARY:
Masquelet's induced membrane technique is a two-stage reconstructive surgery for severe bone fractures commonly used by military orthopedists. The particularity of this technique relies on the synthesis of a biological membrane induced by the transient implantation of a surgical cement (= 1st stage surgery). The presence of the induced membrane in the reconstruction space defines a microenvironment or "biological chamber" favourable to osteogenesis, positively influencing the repair of the lesion after implantation of an autologous bone graft (= 2nd stage of surgery).

In view of the excellent clinical results obtained with this procedure, the Masquelet technique has gradually become a reference treatment in the field of orthopedic and trauma surgery.

However, orthopedic surgeons sometimes observe failures in bone consolidation. To our knowledge, the role played by induced membrane in these therapeutic failures has never been studied.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with traumatic bone loss
* Patient eligible for the induced membrane technique

Exclusion Criteria:

* Patients with post-tumor bone loss
* Patients who are immunocompromised or under immunosuppressive treatment
* Patients with chronic inflammatory disease (diabetes, inflammatory bowel disease)
* Patients with collagenosis
* Patient with a contraindication to sampling
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of patients with traumatic bone loss who are eligible for the induced membrane technique.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Histological profile of induced membrane fragments | Through study completion, an average of 6,5 years
  Presence of abnormalities in the organization of connective fibers. The profile of induced membrane fragments will be compared between patients who respond and patients who do not respond to the induced membrane technique.
Cellular profile of induced membrane fragments | Through study completion, an average of 6,5 years
  Presence of mesenchymal stromal cells, ability of these cells to differentiate into osteoblasts, presence of other cell types (such as adipocytes and osteoclasts).
  The profile of induced membrane fragments will be compared between patients who respond and patients who do not respond to the induced membrane technique.
Secretory profile of induced membrane fragments | Through study completion, an average of 6,5 years
  Determination of proteins secreted by the induced membrane fragments by mass spectrometry or by enzyme-linked immunosorbent assay.
  The profile of induced membrane fragments will be compared between patients who respond and patients who do not respond to the induced membrane technique.
Gene expression profile of induced membrane fragments | Through study completion, an average of 6,5 years
  Expression of several genes of interest related to angiogenesis, mesenchymal stromal cells mobilization, bone formation or resorption and extracellular matrix remodeling.
  The profile of induced membrane fragments will be compared between patients who respond and patients who do not respond to the induced membrane technique.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital d'Instruction des Armées Percy, Clamart
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé

IPD SHARING:
Plan to Share IPD: Undecided